CLINICAL TRIAL: NCT02238769
Title: Diagnostic Accuracy of 18F-FluoroethylCholine Positron Emission Tomography for Hepatocellular Carcinoma
Brief Title: 18F-FluoroethylCholine Positron Emission Tomography: a Promising Diagnostic Tool for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FECH-PET-2014
Record Dates: First submitted 2014-09-03; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma, 18F-FluoroethylCholine PET
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatocellular Carcinoma: 18F-FluoroethylCholine PET will show the difference between HCC lesions and normal liver tissue
  Interventions: Device: 18F-FluoroethylCholine PET

INTERVENTIONS:
Device: 18F-FluoroethylCholine PET — 18F-FluoroethylCholine PET will be performed before any treatment of patients. 18F-FECH was prepared and provided by Nuclear Medical Center of our hospital.PET scan was performed using SIEMENS/CTI（index） EXACT HR（high resolution) +.

SUMMARY:
18F-FluoroethylCholine (18F-FECH) is a new tracer used in PET synthesized by Nuclear Medical Center of Peking Union Medical College Hospital and is favored for diagnosis of primary brain tumor. Although 18F-FECH showed a high presence of biological distribution in liver, 18F-FECH PET may have a higher sensitivity in diagnosis of intra- and extra-hepatic lesions of HCC respectively than those of 18F-FDG or 11C-acetate PET scan, and 18F-FECH PET could be a promising tool in diagnosis and staging, therapy selection and prognostic evaluation for HCC patients. However, much more cases are required to verify this theory. The purpose for this study is to establish the model of clinical experimental prospective study, and to evaluate the sensitivity, specificity and accuracy of 18F-FECH PET in diagnosis of HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) ranks sixth in cancer incidence and third in cancer mortality worldwide. The diagnosis of HCC is made on the basis of tumor markers and imaging examination such as CT or MRI at present. The most commonly used serological marker is alpha-fetoprotein (AFP), of which the sensitivity ranges from 33% to 85% and is only 56.3% on average. The sensitivities of CT and MRI in the diagnosis of small HCC lesions (diameter ≤ 2cm) reported to be about only 20% and 27% respectively. Therefore, distinction from small malignancies to benign lesions by using tumor marker tests or conventional imaging method may be difficult and unreliable.

Positron emission tomography (PET) is widely used in oncology. Fluorine-18-Fluorodeoxyglucose (18F-FDG) PET seems to be a powerful imaging method in diagnosis of breast cancer, gastric cancer, and colorectal cancer. However, our previous study has showed the limited diagnostic sensitivity of 18F-FDG PET in HCC lesions (54%), which makes 18F-FDG PET of no additional value to conventional imaging in the diagnosis of HCC. 11C-acetate PET has been used in the diagnosis of various malignant tumors. Compared with 18F-FDG PET, 11C-acetate PET has an increased sensitivity (63.6%) in diagnosis of well-differentiated HCC, which presents a high avidity for acetate rather than glucose. However, it still has a high rate of misdiagnoses, and has been insufficient to complement 18F-FDG PET for a better diagnosis.

18F-FECH is a new tracer used in PET synthesized by Nuclear Medical Center of Peking Union Medical College Hospital and is favored for diagnosis of primary brain tumor. 18F-FECH showed a high presence of biological distribution in liver and was rarely used in HCC diagnosis. Recently, we find that 18F-FECH may presents a higher sensitivity in diagnosis of intra- and extra-hepatic lesions of HCC respectively, which are much higher than those of 18F-FDG or 11C-acetate PET scan. Therefore, 18F-FECH PET could be a promising tool in diagnosis and staging, therapy selection and prognostic evaluation for HCC patients. However, more researches are required to assess the accuracy and application prospect of 18F-FECH PET in the diagnosis of HCC.

The aim of our study are:

1. To establish the model of clinical experimental prospective study, and to evaluate the sensitivity, specificity and accuracy of 18F-FECH PET in diagnosis of HCC.
2. To assess the accuracy of 18F-FECH PET in diagnosis of HCC at the early stage (diameter ≤ 3cm), and to explore the difference of 18F-FECH PET imaging findings between early or late HCC lesions in order to guide the clinical application in the future.
3. To evaluate the effectiveness of 18F-FECH PET in differential diagnosis of HCC and liver benign lesions such as hemangioma, focal nodular hyperplasia (FNH), hepatic adenoma, and primary neuroendocrine tumors.
4. To evaluate the effectiveness of 18F-FECH PET in differential diagnosis of HCC and other hepatic malignancies (ICC, HCC-ICC, CC, malignant lymphadenoma, sarcoma or adenocarcinoma) or metastatic neoplasm.
5. To explore the clinical pathological characteristics of HCC patients which may affect the accuracy of 18F-FECH PET in diagnosis of HCC, and to determine under which conditions the patients are suitable for 18F-FECH PET scan and to explore whether the liver disease itself, such as cirrhosis would affect the diagnostic efficacy of 18F-FECH PET. The characteristics include tumor size (diameter ≤ or > 3cm), number of lesions, Edmondson grade (including immuno-histochemistry), tumor thrombus in portal vein, extra-hepatic metastasis, clinical stage; patients' age, sex, history of disease (including chronic hepatitis, cirrhosis, metabolic disease such as hepatolenticular degeneration, genetic diseases such as Gaucher disease and Niemann-Peak disease), liver function (Child-Pugh grade) and coagulation function.
6. To search the differences of accuracy between 18F-FECH PET and 18F-FDG PET in diagnosis of HCC, and to explore the value of them in HCC diagnosis.
7. To detect the relationship between 18F-FECH PET imaging findings and the prognosis of HCC patients under the same treatment, and to determine whether the 18F-FECH PET imaging findings can be used as independent factors in evaluating prognosis of HCC.
8. To explore the mechanism of imaging features and specific findings of 18F-FECH PET in the diagnosis of HCC, which may offer potential help for analyzing 18F-FECH PET results.

ELIGIBILITY:
Inclusion Criteria:

1. patients should be older than 18 years;
2. patients were preliminary diagnosed as HCC by conventional imaging examinations such as enhanced CT or MRI, or by history of liver disease or tumor marker texts (AFP, CA19-9);
3. the final diagnosis should be based on pathological results.

Exclusion Criteria:

1. women during pregnant stage or breast-feed stage;
2. patients suffered from serious neurological or psychiatric diseases so that (such as claustrophobia) cannot rest for 15~30 min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The studied population is consisted of the patients with a suspicion of HCC treated in our hospital from September 2014 to August 2015.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
SUVratio of FECH PET | 1 year
  The studied population will be consisted of the patients with a suspicion of HCC treated in our hospital from October 2014 to October 2015. Patients following the Inclusion criteria and Exclusion criteria will undergo 18F-FECH and 18F-FDG PET examinations before clinical treatments. The maximum standard uptake value (SUVmax) of liver lesions and the mean SUV of the non-affected liver (SUVmean) will be measured. SUVratio will be calculated as SUVmax/ SUVmean.

SECONDARY OUTCOMES:
Patients' lifespan | 2 years
  Patients' lifespan and survival condition will be measured. The follow-up of the patients will end in April 2017. Tumor size, intensity of arterial enhancement on dynamic imaging of the primary lesion, and extent of disease after patients' treatments will be measured on CT and/or MRI.

OTHER OUTCOMES:
Data analysis | 2 months
  A receiver operating characteristic (ROC) curve will be performed to assess the cutoff for the SUV. Sensitivity and specificity are based on McNemar's test. The results of 18F-FECH PET and pathological diagnosis for matching are compared by Kappa test. Pearson's chi square and Fisher's exact correlation tests are used for categorical data analyses. Survival analysis will be performed and survival curves were plotted by Kaplan-Meier method. Log-rank test is used for the comparison between the two survival curves. One-way ANOVA with Tukey's test is used to evaluate the gene expressions. Date analysis will help us to evaluate the sensitivity, specificity and accuracy of 18F-FECH PET in diagnosis of HCC, to assess the accuracy of 18F-FECH PET in diagnosis of HCC at the early stage (diameter ≤ 3cm), and to explore the difference of 18F-FECH PET imaging findings between early or late HCC lesions in order to guide the clinical application in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Yilei Mao, MD, Principal Investigator — PUMCH
Locations (1):
- Department of liver surgery; Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Huo L, Dang Y, Lv J, Xing H, Li F. Application of dual phase imaging of 11C-acetate positron emission tomography on differential diagnosis of small hepatic lesions. PLoS One. 2014 May 9;9(5):e96517. doi: 10.1371/journal.pone.0096517. eCollection 2014. PMID 24816814
- [Background] Mao Y, Yang H, Xu H, Lu X, Sang X, Du S, Zhao H, Chen W, Xu Y, Chi T, Yang Z, Cai J, Li H, Chen J, Zhong S, Mohanti SR, Lopez-Soler R, Millis JM, Huang J, Zhang H. Golgi protein 73 (GOLPH2) is a valuable serum marker for hepatocellular carcinoma. Gut. 2010 Dec;59(12):1687-93. doi: 10.1136/gut.2010.214916. Epub 2010 Sep 28. PMID 20876776
- [Background] Larsson P, Arvidsson D, Bjornstedt M, Isaksson B, Jersenius U, Motarjemi H, Jacobsson H. Adding 11C-acetate to 18F-FDG at PET Examination Has an Incremental Value in the Diagnosis of Hepatocellular Carcinoma. Mol Imaging Radionucl Ther. 2012 Apr;21(1):6-12. doi: 10.4274/Mirt.87. Epub 2012 Apr 1. PMID 23487415